CLINICAL TRIAL: NCT03982264
Title: Cap Endoscopic Mucosal Resection(EMR-C) Versus Endoscopic Submucosal Dissection(ESD) for Treatment of Rectal Neuroendocrine Tumor(NET) Less Than 10mm
Brief Title: Endoscopic Treatment of Rectal Neuroendocrine Tumor(NET) Less Than 10mm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2017-077
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Rectal Neuroendocrine Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD group (Active Comparator): In ESD group, enrolled patients will receive the treatment modality of ESD to remove the rectal NET
  Interventions: Procedure: ESD procedure
- EMR-C group (Experimental): In EMR-C group, enrolled patients will receive the treatment modality of EMR-C to remove the rectal NET
  Interventions: Procedure: EMR-C procedure

INTERVENTIONS:
Procedure: ESD procedure — ESD were all performed as the standard procedure that has been widely described and used. A diluted sodium hyaluronate solution was injected submucosally. Mucosal incision and submucosal dissection were performed by using either Hook knife (Olympus Medical, Japan) or a dual-knife (Olympus Medical, Japan) . After the resection was finished, all of the visible vessels on the artificial ulcer bed were thoroughly coagulated with argon plasma coagulation to prevent postoperative bleeding.
  Arms: ESD group
Procedure: EMR-C procedure — A transparent cap (MH-593; Olympus) was attached to the forward-viewing endoscope. After the endoscope was inserted to the rectum, the snare passed through the sheath and was looped along the inner lip of the cap. The tumor was then suctioned into the cap and the snare was pushed off and closed. After confirming the appropriate snare placement, both the tumor and the overlying mucosa were resected by electric cautery (Endocut Q, effect 2, VIO 200D; ERBE, Tübingen, Germany), and then the removed tumor was sent for pathological examination. Endoscopic examination then was repeated without the transparent cap in order to evaluate the wound carefully in case there was any perforation or bleeding and to ensure the absence of the residual tumor tissues. If there was spurting bleeding or active bleeding, hot forceps were usually to stop the bleeding.
  Arms: EMR-C group

SUMMARY:
Cap-assisted endoscopic mucosal resection (EMR-C) and endoscopic submucosal dissection (ESD) have both been reported to be effective treatment methods for small rectal neuroendocrine tumor (NET) in limited studies. Which one is better has not been determined. We aimed to compare the efficacy and safety of EMR-C and ESD for the treatment of small rectal NET.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years;
* Definite diagnosis of rectal NET less than 10mm;
* Patients plan to receive either EMR-C or ESD treatment.

Exclusion Criteria:

* Serious comorbid diseases such as advanced malignant tumor and organ failure;
* Patients received conventional EMR, snare electrotomy and no treatment;
* Rectal NET with metastasis;
* Pregnant patient;
* Poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
complete resection rate(R0 rate) | within 14 days after procedure
  Complete resection was defined as negative horizontal and vertical margins of specimen.

SECONDARY OUTCOMES:
operating time | intraoperative
  the time from endoscope in to endoscope out
complications rate | within 14 days after procedure
  Complications were defined as perforation or hemorrhage during or after operation.
length of stay | within 14 days after procedure
  calculated from the day of admission to day of discharge
hospitalization cost | within 14 days after procedure
  represent the hospital's costs of being hospitalized
recurrence rate | one year after procedure
  a new rectal NET recurred confirmed by endoscopy and EUS

REFERENCES:
- [Derived] Gao X, Huang S, Wang Y, Peng Q, Li W, Zou Y, Han Z, Cai J, Luo Y, Ye Y, Li A, Bai Y, Chen Y, Liu S, Li Y. Modified Cap-Assisted Endoscopic Mucosal Resection Versus Endoscopic Submucosal Dissection for the Treatment of Rectal Neuroendocrine Tumors </=10 mm: A Randomized Noninferiority Trial. Am J Gastroenterol. 2022 Dec 1;117(12):1982-1989. doi: 10.14309/ajg.0000000000001914. Epub 2022 Aug 23. PMID 36455222